CLINICAL TRIAL: NCT02620254
Title: Mast Cell Connect: A Registry for Patients With Mastocytosis
Status: Completed | Type: Observational
Sponsor: Blueprint Medicines Corporation (Industry)
Collaborators: PatientCrossroads (Industry)
Responsible Party: Sponsor
Other Study IDs: Mastocytosis Registry
Record Dates: First submitted 2015-11-19; First posted 2015-12-02 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Mastocytosis
Keywords: mastocytosis; cutaneous mastocytosis; urticaria pigmentosa; telangiectasia macularis eruptiva perstans (TMEP); diffuse cutaneous mastocytosis; solitary cutaneous mastocytosis; systemic mastocytosis; indolent systemic mastocytosis; smoldering systemic mastocytosis; aggressive systemic mastocytosis; systemic mastocytosis with associated clonal hematologic non-mast cell lineage disease; mast cell leukemia
MeSH Terms: conditions — Mastocytosis; Mastocytosis, Cutaneous; Urticaria Pigmentosa; Telangiectasia macularis eruptiva perstans; Mastocytosis, Systemic; Leukemia, Mast-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years

SUMMARY:
The Mast Cell Connect Registry is a voluntary, observational database that will capture demographic, socioeconomic, and disease information directly from patients with mastocytosis via a secure web-based tool. No experimental intervention is involved.

DETAILED DESCRIPTION:
Mastocytosis is an extremely rare and heterogeneous spectrum of diseases characterized by the buildup of genetically altered mast cells. Patients experience a wide range of symptoms and in some cases, mast cell buildup can lead to organ dysfunction and failure. Current treatments address disease symptoms and not the underlying cause. To facilitate the development of new therapies for mastocytosis, it is important for the community to support clinical trials and to document the impact of the disease, including disease natural history and the impact on patients, in a systematic way. Mast Cell Connect is a web-based registry that allows mastocytosis patients and caregivers to enter information about the experience of the patient living with mastocytosis directly into an online data collection tool.

The Mast Cell Connect Registry allows mastocytosis patients and caregivers to enter information about the experience of the patient living with mastocytosis directly into a web-based data collection tool. Two forms of data will be collected: responses to surveys administered on the web-based portal, and de-identified data curated from medical reports uploaded by patients or their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a diagnosis of mastocytosis, including systemic mastocytosis and cutaneous mastocytosis and any subtypes of these diseases, who is willing and able to provide written online informed consent

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of mastocytosis, including systemic mastocytosis and cutaneous mastocytosis and any subtypes of these diseases.
Sampling Method: Non-Probability Sample
Enrollment: 743 (Actual)
Dates: Start 2015-11; Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Further the understanding of the epidemiology of mastocytosis and its subtypes | Through completion of the study

OTHER OUTCOMES:
Improve the collective understanding of the natural history of mastocytosis and its impact on patients | Through completion of the study
Assist in the development of mastocytosis therapy by increasing participation in clinical trials and other research studies for patients with mastocytosis | Through completion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Anthony L Boral, MD, PhD, Principal Investigator — Blueprint Medicines Corporation
Locations (1):
- Registry participation is worldwide and not limited to this facility, Cambridge, Massachusetts, United States

REFERENCES:
- See also: Related Info — http://www.mastcellconnect.org